CLINICAL TRIAL: NCT04983459
Title: Positron Emission Tomography/Computed Tomography With Prostate Specific Membrane Antigen Ligands for Occult Biochemical Recurrence Detection in Patients With Prostate Cancer: a Single Centre Experience
Brief Title: PSMA PET/CT for Biochemical Recurrence Detection in Patients With Prostate Cancer
Acronym: RB-PSMA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RB-PSMA (29BRC21.0040)
Record Dates: First submitted 2021-06-17; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Prostatic Neoplasms; Recurrence
Keywords: PSMA PET/CT
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate PSMA-PET for the detection of occult biological recurrence in patients with prostatic cancer referred to the Brest University Hospital.

DETAILED DESCRIPTION:
In France, prostate cancer is the most common cancer in men over 50 years of age (nearly 50,000 new cases per year) and is the third leading cause of cancer-related death in men (approximately 9,000 deaths per year).

Among patients who have undergone a curative treatment strategy for localized prostate cancer, between 27% and 53% of them will have a biochemical recurrence within 10 years.

Biochemical recurrence is defined as :

* After total prostatectomy by the persistence of a detectable PSA or the reappearance of a detectable PSA above 0.2 ng/ml after a more or less long period of undetectability.
* After conservative treatment (radiotherapy or brachytherapy) by an increase in PSA above a threshold set at nadir +2 ng/ml Biological recurrence precedes the occurrence of symptomatic metastases by an average of 7-8 years.

Currently, after prostatectomy, when the PSA is < 1 ng/mL, no imaging test is recommended for the assessment of recurrence (grade A recommendation).

The sensitivity of currently available tests does not provide sufficiently discriminating information for this PSA value.

Multiparametric MRI performs well in detecting local recurrence, particularly in the case of PSA > 1 ng/mL (sensitivity of 98%, specificity of 94% for the detection of 5 mm lesions).

18F-choline positron emission tomography (PET-choline) is of interest in the detection of distant lymph node and/or visceral recurrences; indeed, PET-choline has proven its superiority in detection compared with conventional examinations, particularly for PSA values above 2ng/ml with a detection rate of up to 90%.

However, the performance of this examination remains dependent on the PSA level and is low when the PSA level is below 1 ng/ml (sensitivity around 5-24% for a PSA below 1 ng/ml).

The performance of PET-choline is optimised for low PSA by taking into account the PSA doubling time and velocity.

Recently, prostate specific membrane antigen ligand positron emission tomography (PET-PSMA) has emerged as the most promising new molecular imaging modality for the management of prostate cancer.

Prostate-specific membrane antigen (PSMA) is a transmembrane glycoprotein selectively overexpressed in 90-100% of prostate cancer lesions, as well as in metastatic lymph nodes and bone metastases, making it an ideal target for molecular imaging of prostate cancer.

This tracer appears to perform better than other imaging modalities, particularly for low PSA values, with a detection rate of 50% for a PSA level below 0.5 ng/ml compared to 5-20% with PET-choline. Indeed, a 2019 meta-analysis evaluating the value of PSMA-PET in patients with biologic recurrence of prostate adenocarcinoma reported detection rates of 45%, 59%, 75% and 95% for PSA levels < 0.5 ng/mL, between 0.5 and 0.9 ng/mL, between 1 and 1.9 ng/mL and 2 ng/mL respectively.

The aim of this study is to evaluate PSMA ligand PET for the detection of occult biological recurrence in patients with prostatic neoplasia referred to the Brest University Hospital .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or older
* Patients referred for a PSMA PET/CT for biochemical recurrence in the nuclear medicine department of Brest University Hospital

Exclusion Criteria:

* Patients for whom PET-PSMA was performed for other reasons.
* Patient's refusal to have their data used for clinical research purposes

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to the nuclear medicine department of Brest University Hospital for a biological recurrence of a prostatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Detection rate per patient of PET-PSMA for the detection of biochemical recurrence. | 12 months
  To evaluate the detection rate per patient of PET-PSMA for the detection of biochemical recurrence

SECONDARY OUTCOMES:
Detection rate per region of PSMA-PET for the detection of biochemical recurrence | 12 months
  To assess the detection rate per region (prostatic bed, pelvic lymph node, extra pelvic lymph node and distant of PSMA-PET for the detection of biochemical recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Richard Pougnet, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning six months and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.